CLINICAL TRIAL: NCT04927962
Title: Psycho-social Impact of Amelogenesis and Dentinogenesis Imperfecta in Young People
Brief Title: Psycho-social Impact of Amelogenesis and Dentinogenesis Imperfecta
Acronym: AiDiBull
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0255
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Dentinogenesis Imperfecta; Amelogenesis Imperfecta
Keywords: Amelogenesis imperfecta; Dentinogenesis imperfecta; Bullying; Oral health related quality of life; Dental anxiety
MeSH Terms: conditions — Dentinogenesis Imperfecta; Amelogenesis Imperfecta; Bullying | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaires — For youth: self-reported questionnaires (on oral quality of life, bullying and cyberbullying, dental anxiety) and routine clinical examination for adolescents. For one parent: self-reported questionnaires (on perceived oral quality of life of their child and on their own dental anxiety).

SUMMARY:
The purpose of this research is to study the impact of dentinogenesis (DI) and amelogenesis (AI) imperfecta on oral quality of life, exposure to bullying and dental anxiety in a population of adolescents. WThe present study will use validated scales to evaluate the impact of bullying on the oral quality of live of youth aged 10 to 18 years, with non-syndromic DI or AI treated in seven national competence or reference centers in rare oral diseases.

ELIGIBILITY:
Inclusion Criteria:

* be between 10 and 18 years of age,
* consult for a care or follow-up consultation
* having a non-syndromic amelogenesis imperfecta or dentinogenesis imperfecta
* having access to a cell phone and/or tablet and/or personal or family computer
* covered by the social security of one of his parents
* understand French and one of whose parents (or legal representative) understands French
* have declared his or her non-opposition and one of whose parents (or legal representative) has declared his or her non-opposition to participate in the study.

Exclusion Criteria:

* Child presenting for diagnostic consultation and child who cannot read or whose 2 parents (legal representatives) cannot read

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients having a non-syndromic amelogenesis imperfecta or dentinogenesis imperfecta and consulting for a care or follow-up consultation.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Child Oral Health Impact Profile (COHIP) | Baseline
  Difference between the average total COHIP questionnaire score of bullied and non bullied patients at D0 (no follow up is planned). A youth is considered bullied if he or she answers "three or more" at least once on the Bullying and Cyberbullying scale for Adolescent questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VAYSSE, Principal Investigator — University hospital of Toulouse
Locations (7):
- France (7):
  - CHU de Bordeaux, Bordeaux
  - Hospices Civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHU de Nantes, Nantes
  - AP-HP, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - University hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No